CLINICAL TRIAL: NCT01185535
Title: Effects of Topical Anesthesia With Pressure Nebulized 2% Lidocaine During Awake Intubation
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Guangdong Science Committee, Guangdong Science Committee
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20081110362101197410300047
Record Dates: First submitted 2010-07-26; First posted 2010-08-20 (Estimated); Last update posted 2010-08-20 (Estimated); Status verified 2010-04

CONDITIONS: Difficult Airway
Keywords: topical anesthesia; tracheal intubation; difficult airway
MeSH Terms: interventions — Anesthesia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 2 times topical anesthesia for glottis (Active Comparator)
  Interventions: Procedure: times of topical anesthesia for glottis
- 3 times topical anesthesia for glottis (Active Comparator)
  Interventions: Procedure: times of topical anesthesia for glottis
- 4 times topical anesthesia for glottis (Active Comparator)
  Interventions: Procedure: times of topical anesthesia for glottis

INTERVENTIONS:
Procedure: times of topical anesthesia for glottis — topical anesthesia with pressure nebulized 2% lidocaine for glottis either two times or three times or four times
  Other Names: topical anesthesia

SUMMARY:
As reported, about 0.43% patients can not be intubated unevenly because of difficult airway and 30% of the total death of anesthesia due to failed intubation. The difficult airway will disturb the clinical treatment and even threaten the patients' life. But the present methods for tracheal intubation during awake intubation can not provided ideal intubation condition. In this study, the investigators will perform topical anesthesia with the nebulized 2% lidocaine at 10L/min oxygen flow rate, and the observer's assessment of alert and sedation (OAA/S) scale was controlled to 3-4 points by intravenous midazolam,propofol, and remifentanil. Tracheal intubation was performed after topical anesthesia. The arterial pressure (MAP), heart rate (HR) and pulse oxygen saturation (SpO2) were recorded and blood samples were taken to measure stress factor during intubation period.Intubation condition score was assessed and the complications like local anesthetic toxicity, mucosa injury, respiration depress were also recorded. Patients were asked whether they could recall the events during intubation 24 hr after operation. The investigators aim is to evaluate the effect of topical anesthesia with lidocaine nebulized by 10L/min oxygen flow rate during awake tracheal intubation.

DETAILED DESCRIPTION:
90 adult patients for elective surgery under general anesthesia, aged 18-60 years old, Mallampti Ⅰ-Ⅱ class, , were randomly allocated to receive topical anesthesia with pressure nebulized 2% lidocaine for glottis either two times or three times or four times(each group n=30). Before topical anesthesia, the observer's assessment of alert and sedation (OAA/S) scale was controlled to 3-4 points by intravenous midazolam (0.03mg/kg), propofol (2mg/kg/h) and remifentanil (0.05μg/kg/min). Ten minutes after sedation, topical anesthesia was performed with the nebulized 2% lidocaine at 10L/min oxygen flow rate, meantime patients were told to breathe deeply. Tracheal intubation was performed after topical anesthesia. The arterial pressure (MAP), heart rate (HR) and pulse oxygen saturation (SpO2) were recorded and blood samples were taken to measure the serum cortisol and insulin concentration during intubation period. Intubation condition score was assessed and the complications like local anesthetic toxicity, mucosa injury, respiration depress were also recorded. Patients were asked whether they could recall the events during intubation 24 hr after operation.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients aged 18-60 years old with Mallampti Ⅰ-Ⅱ class

Exclusion Criteria:

* Patients who have allergic reaction to the drugs used during anesthesia
* Patients who have a history of gastro-esophageal regurgitation, or with full stomach
* Patients with abnormality of cardiopulmonary function, renal and liver function
* Patients with abnormality of endocrine function
* Patients with increased intracranial pressure or epilepsy

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2010-01; Primary Completion 2010-08 (Estimated); Study Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
Intubation condition score during awake intubation period | one years
  Intubating condition score (Jaw relaxation; Laryngoscopy insertion; Vocal cord position; Coughing; Limb movement; Cuff response)

SECONDARY OUTCOMES:
Stress factor during intubation period | one year
  Blood samples were drawn to measure the serum cortisol and insulin concentration.
Life signs during intubation period | one year
  The arterial pressure (MAP), heart rate (HR) and pulse oxygen saturation (SpO2) were recorded.
The complications during intubation period | one year
  The complications like local anesthetic toxicity, mucosa injury, respiration depress were also recorded. Patients were asked whether they could recall the events during intubation 24 hr after operation.

CONTACTS AND LOCATIONS:
Overall Officials: Jin s qing, doctor, Study Director — Sixth Affiliated Hospital, Sun Yat-sen University
Locations (1):
- lab of The Sixth Affiliated Hospital, Sun Yat-sen University, Guangzhou, Guangdong, China

REFERENCES:
- [Derived] Jiang H, Miao HS, Jin SQ, Chen LH, Tian JL. A pilot study of the effect of pressure-driven lidocaine spray on airway topical anesthesia for conscious sedation intubation. Chin Med J (Engl). 2011 Dec;124(23):3997-4001. PMID 22340331
- See also: PUMED — http://www.ncbi.nlm.nih.gov/sites/entrez